CLINICAL TRIAL: NCT05749432
Title: A Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Antitumor Efficacy of Hemay181 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study of Hemay181 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM181ST1S01
Record Dates: First submitted 2023-02-15; First posted 2023-03-01 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemay181 (Experimental): Part one: Dose Escalation Group Hemay181 will be injected in doses of 4.5 mg/m^2, 9.0 mg/m^2, and 18 mg/m^2 until any drug-related toxicity of grade 2 or higher is observed in any dose group. Next, Hemay181 will be injected in doses of 36mg/m^2, 60mg/m^2, 90mg/m^2, 120mg/m^2, 150mg/m^2, 180mg/m^2, 210mg/m^2 until there are two cases of dose-limiting toxicity in a dose group.
  Part two: Extension Group Hemay181 will be injected in the highest three dose groups that had been assessed until disease progression.
  Interventions: Drug: Hemay181

INTERVENTIONS:
Drug: Hemay181 — Hemay181 will be given intravenously on the first day per cycle, and the treatment cycle is 21-days.

SUMMARY:
The study will be conducted in about 51 participants in total. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetic profile and preliminary antitumor efficacy of Hemay181 in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The primary purpose of this study is to evaluate the safety and tolerability of Hemay181 in patients with advanced solid tumors, and to explore the maximum tolerated dose. The secondary purpose is to evaluate the pharmacokinetic profile of Hemay181 in patients with advanced solid tumors and to evaluate the preliminary evaluation of the anti-tumor efficacy of Hemay181.

The study will be conducted in two parts. Part one, trial will be conducted in about 24 subjects to determine safety and tolerability of Hemay181 in patients with advanced solid tumors. Part two, approximately 15-27 additional subjects with advanced solid tumors are included to better define the tolerability and preliminary efficacy of Hemay181.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 65 years;
2. Subjects must give informed consent to the study before the study entry and voluntarily sign a written informed consent form;
3. Advanced solid tumors patients that confirmed by pathology (histology or cytology) with adequate standard therapy failure or currently have no effective standard treatment (such as breast, liver, lung, gastric cancer, colorectal cancer, etc.); Standard therapy failure is defined as: patients who have undergone at least 2 lines of standard antineoplastic therapy after recurrence/metastasis (including treatment-naïve stage IV) (if only 1-line therapy is recommended for the tumor, standard 1-line therapy shall prevail), and who have been confirmed by the investigator or have a clear disease progression or are intolerable by the medical history;
4. At least one lesion that can be evaluated by CT/MRI (measurable lesions are required) and meet the reproducible evaluation requirements in RECIST V1.1;
5. At least 4 weeks after the latest treatment (chemotherapy, targeted therapy, immunotherapy, radiotherapy, and/or major surgery, etc.), at least 2 weeks after endocrine therapy, and have recovered from the toxic effects caused by previous treatment to lower than grade 1 (CTCAE version 5.0) [patients with hair loss (any grade), pigmentation (any grade), peripheral sensory neuropathy (grade ≤2) can be enrolled];
6. Eastern Cooperative Oncology Group(ECOG) score of 0,1；
7. Life expectancy of at least three months;
8. Adequate bone marrow, liver, kidney function, meeting the following criteria:

   ANC≥1.5×10^9/L, HB≥90g/L, PLT≥75×10^9/L; ALT≤2.5×ULN, AST≤2.5×ULN with no liver metastasis, or ALT≤5×ULN, AST≤5×ULN with liver metastasis; TBIL≤1.5×ULN; Serum creatinine ≤1.5×ULN；
9. All female and male subjects must agree and commit to the use of a reliable contraceptive regimen for the duration of the study and for at least 12 weeks after at the last dose of test article.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients with known central nervous system metastatic disease;
3. Positive blood for human immunodeficiency virus (HIV antibody); Positive hepatitis B surface antigen and Hepatitis B virus deoxyribonucleic acid (HBV-DNA)>upper limit of normal; Active hepatitis C virus (HCV) infection;
4. Patients with active infection requiring intravenous anti-infective therapy;
5. Patients with a history of irinotecan allergic reactions or previous irinotecan gastrointestinal toxicity ≥ grade 3;
6. Have received drug therapy from other clinical trials within 4 weeks prior to enrollment;
7. Known allergy to the active ingredient or excipients of the test drug;
8. The investigator believes that the subject has any clinical or laboratory abnormalities and is not suitable to participate in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 3 weeks of treatment
Incidence of dose-limiting toxicity (DLT) in each dose group | 3 weeks of treatment
Maximum tolerated dose (MTD) or Maximum climbing dose (MAD) of Hemay181 | 3 weeks of treatment
Subsequent recommended doses of Hemay181 | 3 weeks of treatment

SECONDARY OUTCOMES:
Objective Response Rate | 3 weeks of treatment
Duration of Response | 3 weeks of treatment
Disease Control Rate | 3 weeks of treatment
Time to Response | 3 weeks of treatment
Progression-Free Survival | 3 weeks of treatment
Maximum Plasma Concentration （Cmax） | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Time to reach maximum concentration （Tmax） | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Elimination half life(t1/2) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Plasma Clearance（CL) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Mean Residence Time from 0 to last time of quantifiable concentration(MRT 0-t) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Mean Residence Time from 0 to infinite time(MRT 0-∞) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Area under the plasma concentration-time curve from 0 to last time of quantifiable concentration(AUC 0-t) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Area under the plasma concentration-time curve from 0 extrapolated to infinite time(AUC 0-∞) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Percentage of the residual area (AUC%Extra) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Volume of distribution(Vz) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile
Elimination rate constant(λz) | 0，0.75, 1.5, 1.75, 2, 2.5, 3.5, 5.5, 9.5, 13.5, 25.5, 49.5, 73.5, 97.5, 121.5 hours post-dose on day 1, and 0，1.5, 2.5 hours post-dose on day 22
  Pharmacokinetic (PK) profile

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China